CLINICAL TRIAL: NCT05416385
Title: Combining Intraplaque Neovascularization With Risk Stratification by Carotid Stress ECHO
Brief Title: Carotid Intraplaque Neovascularization Combined With Stress Echo
Acronym: CIRCE
Status: Recruiting | Type: Observational
Sponsor: Dr. Amer Johri (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor-Investigator, Dr. Amer Johri, Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: DMED-2469-21-6032717; CG#21007 (Other Grant/Funding Number: Lantheus Medical Imaging, Inc.); 452696 (Other: Canadian Institutes of Health Research)
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Acute Coronary Syndrome; Ischemic Heart Disease; Myocardial Infarction; Carotid Artery Diseases
Keywords: Ultrasound; Echocardiography; Stress Testing; Contrast Enhanced Ultrasound
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Acute Coronary Syndrome; Myocardial Ischemia; Myocardial Infarction; Carotid Artery Diseases | interventions — Contrast Media; perflutren

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cardiac outpatients: Subjects referred for outpatient stress echocardiogram (SE).
  Interventions: Other: Carotid Contrast Enhanced Ultrasound

INTERVENTIONS:
Other: Carotid Contrast Enhanced Ultrasound — Carotid Contrast-Enhanced Ultrasound (CEUS), a diagnostic ultrasound enhancing agent that opacifies the blood to delineate the vessel walls.
  Other Names: Contrast injection, DEFINITY®, Perflutren Lipid Microsphere

SUMMARY:
The root cause of heart attacks and strokes is atherosclerosis, the hardening and thickening of blood vessels due to the presence of "plaque" which is a build-up of fat and cholesterol in the walls of vessels. To diagnose heart disease, patients receive a stress test to find out if they require surgery. Up to 52% of patients receiving an angiogram (surgery) to look at plaque blockages in the heart are found to be normal (no blockage). Patients who are suspected of having heart disease often undergo a stress test, which helps cardiologists decide if the patient has heart disease, but stress tests can give false results. In Ontario alone, 90% are stress tests are found to be normal and patients are sent home with little follow-up. Of these 3-5% (~4,000 patients/year) will have a major cardiovascular event (heart attack, surgery, or death) within 3 years. We need to improve the stress test accuracy to reduce cardiac outcome. We now know that it is not just the total amount of plaque that leads to heart attacks and strokes, but the composition of the plaque that can lead to breakage causing a heart attack. Plaques are soft and fragile, and typically contain fat and small leaky blood vessels within their cores. If we are able to identify patients that have leaky plaques using ultrasound, we may be able to improve the accuracy of stress testing. We propose a study looking at the combination of stress testing (assessing heart function) and neck ultrasound (assessing plaque composition), to identify patients at risk for cardiovascular events (heart attacks and death). We will enrol patients from 6 sites across Canada and follow-them for cardiac outcome for 3 years.

DETAILED DESCRIPTION:
Primary Aim: To determine if carotid intraplaque neovascularization score (IPN) combined with stress echo (SE) [IPN+SE] enhances prediction of 3-year major adverse cardiovascular events (MACE) compared to SE alone.

Objectives: 1) The % change in test sensitivity of IPN+SE for predicting 3-year MACE compared with SE alone. 2) The Net Reclassification Improvement (NRI) for MACE will be determined (patients "missed" by the SE, but captured as high risk for MACE by IPN).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women >18 years;
2. Referred for a clinically indicated SE for assessment of ischemia and risk stratification;
3. Able and willing to give informed consent.

Exclusion Criteria:

1. Emergency procedure, or active acute coronary syndrome (active chest pain, ischemic electrocardiogram changes, or cardiac enzyme elevation);
2. Referral for viability, pulmonary hypertension, or valve assessment;
3. Referral outside of the normal working hours;
4. History of significant CAD: percutaneous coronary intervention (PCI), coronary artery bypass graft (GABG), or coronary angioplasty;
5. History of stroke or myocardial infarction (MI);
6. Known or documented hypersensitivity or allergy to perflutren (DEFINITY® contrast agent);
7. Known or documented allergy to Polyethylene Glycol (Peg) a component of DEFINITY®;
8. History of carotid surgery (endarterectomy or stenting);
9. Any serious medical condition or complication from the stress test that according to the investigator could interfere with the carotid scan or optimal care;
10. Currently pregnant or breastfeeding;
11. Previous enrolment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Low to intermediate risk outpatient subjects referred for stress echo (SE) for assessment of ischemia and risk stratification will be screened for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2026-08-16 (Estimated); Study Completion 2026-08-16 (Estimated)

PRIMARY OUTCOMES:
Our primary outcomes will be the improvement in sensitivity and negative predictive value (NPV). | This is a 5-year study. The outcome follow up for mace will be 3-years from the index date (SE).
  Our primary analysis will compare the sensitivity of an established binary test based on SE alone to a binary test based on SE and plaque assessment (using established thresholds, IPN≥1.25) to predict 3-year MACE.

CONTACTS AND LOCATIONS:
Overall Officials: Amer Johri, MD, Principal Investigator — Queen's University
Locations (6):
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Dalhousie University, Halifax, Nova Scotia
  - The Kingston Heart Clinic, Kingston, Ontario
  - Queen's University, Cardiovascular Imaging Network at Queen's (CINQ), Kingston, Ontario
  - Unity Health Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No